CLINICAL TRIAL: NCT04156191
Title: An Open Label, Phase 1, Pharmacokinetics, Maximal Usage Pharmacokinetics, Safety, and Efficacy Study of ARQ-151 Cream 0.15% or ARQ-151 Cream 0.05% Administered QD in Adolescent and Pediatric Subjects With Mild to Moderate Atopic Dermatitis
Brief Title: Pharmacokinetics (PK), Safety, Efficacy and Maximal Use PK of ARQ-151 in Adolescents/Children With Mild/Moderate Eczema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ-151-105
Record Dates: First submitted 2019-11-03; First posted 2019-11-07 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Atopic Dermatitis (Eczema)
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARQ-151 cream 0.15% or 0.05% (Experimental): Open-label study of 0.15% or 0.05% active concentration
  Interventions: Drug: ARQ-151 cream 0.15%; Drug: ARQ-151 cream 0.05%

INTERVENTIONS:
Drug: ARQ-151 cream 0.15% — ARQ-151 cream 0.15% applied to atopic dermatitis lesions once a day for 28 days
Drug: ARQ-151 cream 0.05% — ARQ-151 cream 0.05% applied to atopic dermatitis lesions once a day for 28 days

SUMMARY:
This is a research study where all subjects will receive study medication to understand how the body processes the study medication, and to determine the PK, safety and efficacy of ARQ-151 cream 0.15% or 0.05% in adolescent and pediatric subjects with mild to moderate AD. At entry, subjects in Cohorts 1-3 will have 1.5-35% Body Surface Area involvement (excluding the scalp, palms, soles) and mild or moderate atopic dermatitis (AD) based on vIGA-AD. Cohort 2 and Cohort 3 will be performed in parallel and may commence after results are available from ARQ-151-212, a Phase 2 study evaluating ARQ-151 cream 0.05% and 0.15% administered once a day for 4 weeks in adolescents and adults with mild to moderate AD affecting 1.5% to 35% BSA.

For the maximal usage PK study (Cohorts 4-8), subjects will have BSA involvement (excluding the scalp, palms, soles) of ≥ 35% in subjects 3 months old to 11 years old (inclusive) or ≥25% in subjects 12 to <17 years old with mild or moderate AD .

Seven groups will be evaluated, including:

* Cohort 1: ARQ-151 cream 0.15% in adolescents (12-17 years old; inclusive)
* Cohort 2: ARQ-151 cream 0.15% in children 6-11 years old (inclusive)
* Cohort 3: ARQ-151 cream 0.15% in children 2-5 years old (inclusive; will be performed in parallel with Cohort 2)
* Cohort 4: ARQ-151 cream 0.15% in adolescents 12 to <17 years old
* Cohort 5: ARQ-151 cream 0.15% in children 6-11 years old (inclusive)
* Cohort 6: ARQ-151 cream 0.15% in children 2-5 years old (inclusive)
* Cohort 7: ARQ-151 cream 0.05% in children 2-5 years old (inclusive)
* Cohort 8: ARQ-151 cream 0.05% in children 3 months old to less than 2 years old

Subjects will apply ARQ-151 cream 0.15% or 0.05% once a day for 28 days to all AD affected areas and any newly appearing AD lesions that arise during the study, except on the scalp.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of parent(s) or legal guardian, and, if age appropriate, assent by the subject, as required by local laws.
2. Males or females, 12-17 years old (inclusive; Cohort 1), or 6-11 years old (inclusive; Cohort 2), or 2-5 years old (inclusive; Cohort 3), and in the maximal usage PK study subjects aged 12 to <17 years old (Cohort 4), 6 to 11 years old (Cohort 5), 2-5 years old (Cohort 6 and Cohort 7), or 3 months to less than 2 years old (Cohort 8).
3. Clinical diagnosis of active atopic dermatitis for at least 3 months (2 weeks for Cohort 8).
4. EASI Score ≥5.
5. vIGA-AD score of 'Mild' ('2') or 'Moderate ('3').
6. Has AD involvement of 1.5 to 35% BSA (Cohorts 1-3) or ≥25% BSA (Cohorts 4-7), all excluding the scalp, palms, soles; or for Cohort 8 ≥35% BSA excluding the scalp, perioral, and below wrists/ankles .
7. Females of childbearing potential must have a negative serum pregnancy test at Screening and, if sexually active, agree to use birth control throughout the trial.
8. In good health as judged by the Investigator, based on medical history, physical examination, and clinical tests.

Exclusion Criteria:

1. Subjects with any serious medical or psychiatric condition or clinically significant physical examination or test abnormality that would prevent study participation or place the subject at significant risk.
2. Subjects with unstable AD or any consistent requirement for high potency topical steroids to manage AD signs or symptoms.
3. Subjects who cannot discontinue the use of strong P-450 cytochrome inducers or inhibitors.
4. Subjects who are unwilling to refrain from prolonged sun exposure and from using a tanning bed or other artificial light emitting devices (LEDs) for 4 weeks prior to Baseline/Visit 2 and during the study.
5. Subjects who cannot discontinue systemic and/or topical therapies.
6. Current or a history of cancer within 5 years with the exception of fully treated skin basal cell carcinoma, cutaneous squamous cell carcinoma or carcinoma in situ of the cervix.
7. Subjects with actively infected AD or any infection that required oral or intravenous administration of antibiotics, antifungal or antiviral agents
8. Known or suspected:

   1. severe renal insufficiency or moderate to severe hepatic disorders (Child-Pugh B or C)
   2. history of chronic infectious disease (e.g., hepatitis B, hepatitis C, or human immunodeficiency virus (HIV))
   3. hypersensitivity to component(s) of the investigational product
   4. history of severe depression, suicidal ideation, Baseline/Screening C-SSRS indicative of suicidal ideation, whether lifetime or recent/current
9. Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
10. Subjects (12 to 17 years old, inclusive) with modified PHQ-A score ≥10 at Screening or Baseline visits.
11. Subjects (6 to 11 years old, inclusive) with a CDI-2 (parent report) raw score >20 at Screening/Baseline
12. Subjects with a history of a major surgery within 4 weeks prior to Baseline/Visit 1 or subjects who have a major surgery planned during the study.
13. Subjects with prior exposure to ARQ-151
14. Subjects 3 to <12 months old who were premature at birth
15. Subject is nursing and subject's mother requires high dose systemic steroids

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of roflumilast and its N-oxide metabolite | 4 weeks
  Maximum observed plasma concentration of drug in plasma
Area under the plasma concentration-time curve within a dosing interval (AUC) for roflumilast and its N-oxide metabolite | 4 weeks
  The area under the plasma concentration-time curve (AUC) is a method of measurement of the total exposure of a drug in plasma.
Treatment Emergent Adverse Events (TEAE) | 4 weeks
  Number of participants with adverse events during treatment will be assessed.

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) Total Score Change and Percent Change in Total Score | Baseline, Week 2, and Week 4
  Change in EASI Total Score at weeks 2 and 4 and percent change from baseline in EASI Total Score at weeks 2 and 4. EASI combines the assessment of the severity of lesions and the area affected into a single total score in the range 0 (no disease) to 72 (maximal disease). To calculate the EASI, the sum of the severity rating (0 to 3 with 3 being the most severe) for four clinical signs are multiplied with the numerical value of the area affected and with the percentage of the four body areas.
Eczema Area and Severity Index Score 100%, 90%, 75%, and 50% Improvement (EASI100, EASI90, EASI75, and EASI50) | Baseline, Week 2, and Week 4
  Proportion of patients with a 100%, 90%, 75%, and 50% or greater improvement in Eczema Area and Severity Index (EASI100, EASI90, EASI75, and EASI50) score from baseline to each study visit. EASI combines the assessment of the severity of lesions and the area affected into a single total score in the range 0 (no disease) to 72 (maximal disease). To calculate the EASI, the sum of the severity rating (0 to 3 with 3 being the most severe) for four clinical signs are multiplied with the numerical value of the area affected and with the percentage of the four body areas.
Achievement of a Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) score of 'clear' or 'almost clear' at each study visit, or 'clear' or 'almost clear' with a 2-point improvement from baseline at each study visit | Baseline, Week 2, Week 4
  The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4 where 0 is clear).
Change from baseline in vIGA-AD score at each study visit | Baseline, Week 2, Week 4
  The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4 where 0 is clear).
Body Surface Area (BSA) Involvement Change | Baseline, Week 2, Week 4
  Change from baseline in BSA involvement at each study visit.
Worse Itch Numerical Rating Score (WI-NRS) Pruritis Score Change | Baseline, Week 2, Week 4
  Change from baseline in WI-NRS pruritus score at each study visit. WI-NRS is a subject-reported severity of itch at its highest intensity during the previous 24-hour period. The scale is from '0 to 10' ("no itch" to "worst imaginable itch").
WI-NRS Pruritus Score Improvement | Baseline, Week 2, Week 4
  ≥4-point improvement from Baseline in WI-NRS pruritus score at each study visit. WI-NRS is a subject-reported severity of itch at its highest intensity during the previous 24-hour period. The scale is from '0 to 10' ("no itch" to "worst imaginable itch").

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (10):
- United States (10):
  - Arcutis Clinical Site 07, Birmingham, Alabama
  - Arcutis Clinical Site 11, Rancho Santa Margarita, California
  - Arcutis Clinical Site 02, Coral Gables, Florida
  - Arcutis Clinical Site 05, Hialeah, Florida
  - Arcutis Clinical Site 13, Miami, Florida
  - Arcutis Clinical Site 01, Mt. Pleasant, South Carolina
  - Arcutis Clinical Site 06, San Antonio, Texas
  - Arcutis Clinical Site 03, Orem, Utah
  - Arcutis Clinical Site 10, West Jordan, Utah
  - Arcutis Clinical Site 12, Spokane, Washington